CLINICAL TRIAL: NCT01073371
Title: Local Anesthetics New Formulations: From Development to Clinical Tests
Brief Title: Anesthetic Efficacy of Liposomal Prilocaine in Maxillary Infiltration Anesthesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Patrícia Maria Wiziack Zago, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 131843/2008-7
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2008-06

CONDITIONS: Dental Anesthesia Efficacy
Keywords: Liposome; Prilocaine; Dental anesthesia
MeSH Terms: interventions — Prilocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- liposome-encapsulated 3% prilocaine (Active Comparator)
  Interventions: Drug: Prilocaine
- 3% plain prilocaine (Active Comparator)
  Interventions: Drug: Prilocaine
- 3% prilocaine with 0,03IU/mL felypressin (Active Comparator)
  Interventions: Drug: Prilocaine

INTERVENTIONS:
Drug: Prilocaine — 1.8mL infiltration of liposome-encapsulated 3% prilocaine, 3% plain prilocaine or 3% prilocaine with 0,03IU/mL felypressin in the buccal sulcus of the maxillary right canine
  Other Names: Citocaína®

SUMMARY:
This blinded randomized, crossover, three period study aim to evaluate the anesthetic efficacy of liposome-encapsulated 3% prilocaine compared to 3% plain prilocaine and 3% prilocaine with 0,03IU/mL felypressin, after 1.8mL infiltration in the buccal sulcus of the maxillary right canine, in 32 volunteers.

ELIGIBILITY:
Inclusion Criteria:

* good health
* no history of allergy to the components of the local anesthetic formulations tested
* maxillary canine, lateral incisor, and first premolar responsible to electric stimulation

Exclusion Criteria:

* intake of any medication that would alter pain perception
* history of trauma or sensitivity, caries, restorations, periodontal disease and endodontic treatment in the maxillary canine, lateral incisor, and first premolar
* systemic disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Anesthesia success, onset and duration of pulpal and gingival anesthesia. | 10 minutes

SECONDARY OUTCOMES:
Injection pain - Visual Analogue Scale | 1 minute after the injections

CONTACTS AND LOCATIONS:
Overall Officials: Eneida de Paula, PhD, Study Director — University of Campinas, Brazil
Locations (1):
- Piracicaba Dental School, Piracicaba, São Paulo, Brazil